CLINICAL TRIAL: NCT04469933
Title: Predictive Factors of Good Results After Primary Descemet's Membrane Endothelial Keratoplasty (DMEK): Retrospective Study About 102 Eyes
Brief Title: Predictive Factors of Good Results After Primary Descemet's Membrane Endothelial Keratoplasty (DMEK)
Acronym: GOODRMEK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-03ObsCHRMT
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Endothelial Corneal Dystrophy
Keywords: Fuchs endothelial corneal dystrophy; central corneal thickness; endothelial cell density; keratometry
MeSH Terms: conditions — Corneal endothelial dystrophy type 2; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim: Identify predictive factors of good results after primary Descemet's Membrane Endothelial Keratoplasty (DMEK) in Fuchs Endothelial Corneal Dystrophy (FECD).

82 patients (102 eyes) with Fuchs Endothelial Corneal Dystrophy (FECD) underwent DMEK between March 2016 and March 2018 were analyzed. Follow-up time was 12 months. The studied prognostic criteria were: pre-operative Central Corneal Thickness (CCT), CCT's delta between pre and D15 post-operatively, anterior mean keratometry, pre-operative endothelial cell density (ECD) and postoperative ECD at 6 and 12 months, pre-operative visual acuity, donors' and recipients' ages, recipients' sex, rebubbling and triple procedure (DMEK combined with cataract surgery).

DETAILED DESCRIPTION:
Aim: Identify predictive factors of good results after primary Descemet's Membrane Endothelial Keratoplasty (DMEK) in Fuchs Endothelial Corneal Dystrophy (FECD).

A monocentric retrospective observational study was realized at the Regional Hospital Center of Metz-Thionville, Mercy Hospital, Metz, France.

102 eyes of 82 patients with Fuchs Endothelial Corneal Dystrophy (FECD) underwent DMEK between March 2016 and March 2018 were analyzed. Follow-up time was 12 months. The studied prognostic criteria were: pre-operative Central Corneal Thickness (CCT), CCT's delta between pre and D15 post-operatively, anterior mean keratometry, pre-operative endothelial cell density (ECD) and postoperative ECD at 6 and 12 months, pre-operative visual acuity, donors' and recipients' ages, recipients' sex, rebubbling and triple procedure (DMEK combined with cataract surgery). Surgery was considered successful when best spectacle corrected visual acuity (BSCVA) was 0.1 logMar or less (≥0.8) 1 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Over 18,
* had advanced FECD associated with visual symptoms and reduced visual acuity .

Exclusion Criteria:

* Prior intraocular surgery other than cataract
* Other indications for DMEK surgeries than FECD,
* Eyes with corneal (except FECD), retinal or optic nerve diseases
* Per-operative difficulties (tear's graft or complicated unfolding graft)
* Primary graft failure (cornea that failed to clear in the presence of an attached graft)
* Secondary graft failure (corneal decompensation after an initial period of a functional graft)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Included patients' were over 18, had advanced FECD associated with visual symptoms and reduced visual acuity
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Pre-operative Central Corneal Thickness (CCT), | day 1
  Pre-operative CCT (μm) measured by an anterior segment optical coherence tomography (AS-OCT; RS-3000; Nidek Co. Ltd, Japan)
Post-operative Central Corneal Thickness (CCT), | Months 12
  Post-operative CCT (μm) measured by an anterior segment optical coherence tomography (AS-OCT; RS-3000; Nidek Co. Ltd, Japan)
CCT's delta | day 15
  CCT's delta (μm) between pre and D15 post-operatively

SECONDARY OUTCOMES:
anterior mean keratometry | day 1
  anterior mean keratometry (calculated by an auto keratometer Visionix Luneau L67, France)
pre-operative endothelial cell density ECD | day1
  pre-operative ECD (using a non-contact specular microscope CEM-530; Nidek Co. Ltd, Japan)
post-operative endothelial cell density (ECD) | 6 months
  post-operative ECD at 6 months (using a non-contact specular microscope CEM-530; Nidek Co. Ltd, Japan)
post-operative endothelial cell density (ECD) | 12 months
  post-operative ECD at 12 months (using a non-contact specular microscope CEM-530; Nidek Co. Ltd, Japan)
pre-operative Visual Acuity | day 1
  pre-operative Visual Acuity (using Monoyer chart and converted it to logMar scale)
donors' and recipients' ages | day 1
  donors' and recipients' ages
recipients' sex | day 1
  recipients' sex
rate of rebubbling | months 6
  the rate of rebubbling %(postoperative graft detachment)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc PERONE, MD, Principal Investigator — CHR Metz Thionville